CLINICAL TRIAL: NCT02976285
Title: Application of a New Polyester Patch in Arthroscopic Massive Rotator Cuff Repair Significantly Improves Clinical Outcome and Tendon Integrity
Brief Title: Polyester Patch in Massive Rotator Cuff Repair Improves Healing
Status: Completed | Type: Observational
Sponsor: Etzel Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: PitchPatch54
Record Dates: First submitted 2016-11-15; First posted 2016-11-29 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Rotator Cuff Tear
Keywords: arthroscopic rotator cuff repair; patch augmentation
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: arthroscopic rotator cuff repair with a polyester patch — Patients were operated under general anesthesia and a supraclavicular nerve block, in a beach-chair position with 80° forward shoulder flexion and traction between 3-5 kg. After washing and draping a standard viewing portal was placed at the dorsal softspot. Further portals included, a lateral, a dorso-lateral, an antero-lateral and an anterior portal. If additional pathologies were present, they were treated simultaneously and mostly involved the long head of the biceps tendon, treated with tenodesis or tenotomy respectively. After a thorough bursectomy, the rupture was fully visualized and thereafter its size was estimated. Following debridement of the footprint, we used a triple row repair and implanted the patch.

SUMMARY:
The purpose of this study was to assess the impact and potential advantage of a novel synthetic patch augmentation in repair of massive rotator cuff (RC) tears, using clinical and radiological approaches. The investigators hypothesized that implanting this patch will improve individual shoulder function, while reducing re-tear rates compared to the current literature.

DETAILED DESCRIPTION:
To evaluate this, patches were implanted into 54 shoulders and prospectively followed up clinically and radiologically.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were age greater 18 years and a RC tear involving at least two tendons, presenting a massive RC-tear as described by Gerber et al.

Exclusion Criteria:

* We excluded patients older than 75, fatty infiltration grade 4 according to Goutallier, re-ruptures of former repairs and cases with severe osteoarthritis.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 54 patients (38 male / 16 female) 54 shoulders (29 right / 25 left) Mean patient age at the time of surgery was 65 years (range 41 - 75).
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2012-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Function assessed with the Constant-Murley-Score | 25 months
Function assessed with the Subjective Shoulder Value | 25 months

SECONDARY OUTCOMES:
Tendon integrity evaluated radiologically | 1-35 months

IPD SHARING:
Plan to Share IPD: No